CLINICAL TRIAL: NCT03326752
Title: Phase 1b Dose Escalation and Dose Expansion Trial of DV281 in Combination With an Approved Anti-PD-1 Inhibitor in Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: Phase 1b DV281 With an Anti-PD-1 Inhibitor in NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DV9-NSC-01
Record Dates: First submitted 2017-10-19; First posted 2017-10-31 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: Cancer; Lung Cancer; NSCLC; Anti-PD-1 inhibitor; Immuno-oncology; Toll-Like Receptor (TLR) agonist
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — DV281; Nebulizers and Vaporizers; Nivolumab

STUDY DESIGN:
Intervention Model Description: * In the Dose Escalation phase of the study, 5 DV281 dose cohorts will be evaluated in combination with an approved anti-PD-1 Inhibitor.
  * The Dose Expansion phase of the study will establish the Recommended Phase 2 Dose of DV281 in combination with an approved anti-PD-1 inhibitor.
Masking Description: N/A - There is no masking in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Dose Escalation Cohort 1-5 (Experimental): Cohort 1-4
  * DV281 - Dose Level 1-5
  * DV281 in combination with nivolumab
  * DV281 is administered via a breath actuated nebulizer
  Interventions: Drug: DV281; Device: Breath Actuated Nebulizer; Drug: Approved Anti-PD-1 Inhibitor
- Dose Expansion (RP2D) (Experimental): 4 Cohorts
  * Preliminary Recommended Phase 2 dosing of DV281 in combination with nivolumab
  * Cohort 1: Non-squamous and non-EGFR/ ALK mutation and progressed on anti-PD-1/L1 therapy
  * Cohort 2: Non-squamous and EGFR/ ALK mutation and progressed on targeted therapy
  * Cohort 3: Squamous and anti-PD-1/ L1 therapy experienced
  * Cohort 4: Squamous and anti-PD-1/L1 therapy naive
  * DV281 is administered via a breath actuated nebulizer.
  Interventions: Device: Breath Actuated Nebulizer; Drug: DV281 (RP2D); Drug: Approved Anti-PD-1 Inhibitor

INTERVENTIONS:
Drug: DV281 — - Dose Escalation will be the preliminary dose finding phase of the study. Subjects will be enrolled to available Dosing Cohorts.
  Arms: Dose Escalation Cohort 1-5
Device: Breath Actuated Nebulizer — Breath-actuated, electronic system designed to aerosolize liquid medication.
  Other Names: Nebulizer
Drug: DV281 (RP2D) — - Dose Expansion will be enrolled into 4 groups based on NSCLC characteristics.
  Arms: Dose Expansion (RP2D)
Drug: Approved Anti-PD-1 Inhibitor — FDA approved Anti-PD-1 Inhibitor
  Other Names: nivolumab

SUMMARY:
This open-label, multicenter, dose-escalation and expansion trial is designed to evaluate the safety and preliminary efficacy of inhaled DV281 in combination with nivolumabfor the treatment of NSCLC and to select a recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
Pre-clinical studies support the proposed dosing schema to be tested and a potential benefit of the combination of inhaled DV281 with nivolumab for subjects with advanced NSCLC. This study (DV9-NSC-01) is designed for establishing an immunologically optimal RP2D for inhaled DV281 in combination with an approved anti-PD-1 inhibitor. This trial, studying the potential to enhance the efficacy of an approved anti-PD-1 inhibitor in subjects with advanced NSCLC, addresses an unmet need for NSCLC patients having tumors that do not respond or do not respond adequately to anti-PD-1 inhibitor monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Have documented histologically or cytologically confirmed advanced NSCLC as the dominant histology.
* If confirmed EGFR or ALK directed testing warrants actionable targeted therapy, must have confirmed disease progression on targeted therapy or cannot tolerate targeted therapy.
* Aged 18 years and older on the day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2 for Dose Escalation phase and ECOG PS 0 to 1 for Dose Expansion phase
* Adequate organ function as indicated by laboratory values
* Life expectancy, in the opinion of the investigator, of at least 3 months

Exclusion Criteria

* Condition of the subjects lung anatomy is such that proper delivery of inhaled DV281 to the specific location of intra-thoracic tumor(s) could be compromised
* Any known additional malignancy that is progressing or required active treatment in the last 3 years
* Current or history of clinically significant non-infectious pneumonitis
* History of clinically severe lung disease, asthma, or chronic obstructive pulmonary disease (COPD) requiring emergency management and/or hospitalization in the last year
* Received more than 30 Gy of conventional radiation therapy in the thoracic region within 26 weeks prior to study enrollment
* Is expected to require any other form of anti-cancer therapy while in the trial. Zoledronic acid or denosumab as supportive care for bone metastases will be allowed if started prior to study enrollment
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10 mg of prednisone or equivalent) or any other form of immunosuppressive therapy (including immune modulators or systemic corticosteroids) that cannot be discontinued safely within 14 days prior to study enrollment
* Has a medical condition that requires immunosuppression
* Active autoimmune disease requiring systemic treatment in the past 2 years or a disease that requires immunosuppressive medication including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Known central nervous system metastases, brain metastases, or carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Dose Escalation | DLT assessment period - Day 1 through Day 28.
  Incidence of dose-limiting toxicities (DLTs)
Dose Expansion | 1 year after last subject is enrolled in the Dose Expansion phase of study
  Objective response rate (ORR) of dosing regimen established during the Dose Escalation
Dose Expansion | 1 year after last subject is enrolled in the Dose Expansion phase of the Study
  Duration of Response (DOR) and time to response.

SECONDARY OUTCOMES:
Dose Escalation | IFN response assessment period - Day 1 through Day 21
  Assess IFN-a induced gene expression in blood when DV281 is administered as a monotherapy and in combination with an approved anti-PD-1 inhibitor
Dose Expansion | 1 year after last subject is enrolled in the Dose Expansion phase of study
  Incidence of treatment related AE's as assessed by CTCAE Version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garon, MD, Principal Investigator — University of California, Los Angeles
Locations (6):
- United States (6):
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Ronald Reagan University of California Los Angeles Medical Center, Santa Monica, California
  - Allina Health, Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No